CLINICAL TRIAL: NCT03262779
Title: A Phase II Study of Combination Immunotherapy With Ipilimumab and Nivolumab in Patients With Advanced Non-small Cell Lung Cancer Resistant to Anti-PD-1-axis Therapy
Brief Title: Ipilimumab and Nivolumab in Patients With Anti-PD-1-axis Therapy-resistant Advanced Non-small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000020343
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab

STUDY DESIGN:
Intervention Model Description: This a phase II study employing a Simon two-stage design. If there is at least one response or prolonged stability (> 24 weeks) using immune related Response Criteria (irRC) appreciated in the first 10 patients who initiate trial therapy, a total of 40 patients will be enrolled. An additional 10 patients with acquired resistance to anti-PD-1 axis therapy will be enrolled in an exploratory cohort receiving the same therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- combination nivolumab and ipilimumab - primary (Experimental): Combination therapy with nivolumab 3 mg/kg administered intravenously (IV) every 2 weeks, and ipilimumab 1 mg/kg administered IV every 6 weeks in patients with primary resistance.
  Interventions: Biological: combination nivolumab and ipilimumab
- combination nivolumab and ipilimumab - acquired (Experimental): Combination therapy with nivolumab 3 mg/kg administered intravenously (IV) every 2 weeks, and ipilimumab 1 mg/kg administered IV every 6 weeks in patients with acquired resistance.
  Interventions: Biological: combination nivolumab and ipilimumab

INTERVENTIONS:
Biological: combination nivolumab and ipilimumab — Combination therapy with nivolumab 3 mg/kg administered intravenously (IV) every 2 weeks, with ipilimumab 1 mg/kg administered IV every 6 weeks.

SUMMARY:
The investigators propose a trial to evaluate if the addition of ipilimumab to nivolumab after primary or acquired resistance to anti- programmed death 1 (PD-1) axis therapy can lead to objective radiographic tumor regression.

DETAILED DESCRIPTION:
Approximately 20 percent of unselected patients with advanced non-small cell lung cancer (NSCLC) and progression during or after standard first line chemotherapy will experience tumor response to nivolumab. Treatment options for patients who are not responsive to programmed death 1 (PD-1) axis inhibitor therapy are limited, and the mechanisms of primary resistance are poorly understood.

The combination of nivolumab and ipilimumab is currently FDA approved for the treatment of advanced melanoma based on superiority to either agent alone5. The results of a phase I study evaluating combination therapy with nivolumab and ipilimumab in patients with advanced NSCLC (NCT01454102) were presented at the annual American Society of Clinical Oncology (ASCO) meeting in 20166. Dosing of nivolumab 3 mg/kg every 2 weeks and ipilimumab 1 mg/kg every 6 weeks yielded an objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 of 39%, with one-year survival rate of 69% and grade 3-4 treatment-related adverse event rate of 33%. These results prompted an ongoing phase III study comparing this regimen to standard first line chemotherapy, nivolumab monotherapy or combination therapy with chemotherapy and nivolumab for patients with advanced NSCLC (NCT02477826).

The investigators propose a trial to evaluate if the addition of ipilimumab to nivolumab after primary resistance to anti-PD-1 axis therapy can lead to objective radiographic tumor regression. It is hypothesized that ipilimumab will enable more effective immune priming in some patients, resulting in the trafficking of tumor-specific cytotoxic T cells to the tumor, as well as depletion of tumor-permissive T regulatory cells. With concurrent nivolumab, PD-1 inhibition in the tumor will enable effective anti-tumor attack by tumor-specific T cells. Serial tumor biopsies and blood collections will allow interrogation of changes in the tumor microenvironment (and periphery) that support this hypothesis.

The investigators will primarily enroll patients who have experienced progression of NSCLC after anti-PD-1- axis therapy without initial response to such therapy ('primary resistance'). A smaller cohort of patients with acquired resistance to anti-PD-1 axis therapy (i.e. progression after initial response) will additionally be accrued.

The study record was updated to add individual arms for those with primary resistance and acquired resistance. The intent of the study is not to compare these treatment arms.

ELIGIBILITY:
Inclusion Criteria

A. Signed Informed Consent B. Ability to comply with the protocol C. Age ≥18 years D. Histologically or cytologically documented, locally advanced or metastatic (i.e., Stage IIIB not eligible for definitive chemoradiotherapy, Stage IV, or recurrent) NSCLC (per the American Joint Committee /AJCC staging system) E. ECOG performance status of 0 to 2 F. Measurable disease, as defined by RECIST v1.1. Previously irradiated lesions can be counted as target lesions if clearly progressing after radiation.

G. Chemotherapy-naive and treated patients will be eligible, with no limit on number of prior therapies. Patients with NSCLC known to harbor an ALK rearrangement, or EGFR mutation known to be sensitive to FDA-approved tyrosine kinase inhibitors (TKI), are only eligible after experiencing disease progression (during or after treatment) or intolerance to an FDA approved EGFR TKI or ALK TKI, respectively.

1. Patients with TKI-treated EGFR mutant NSCLC harboring the secondary EGFR T790M tumor must have received prior osimertinib
2. Patients with crizotinib-treated ALK rearranged NSCLC must have received a next generation ALK inhibitor (e.g. ceritinib, alectinib or brigatinib) H. Prior palliative radiotherapy must have been completed at least 2 weeks before the first dose of study drug.

I. Anti- PD-1 Axis therapy (anti-PD-1 or anti-PD-L1, e.g. nivolumab, pembrolizumab, atezolizumab, durvalumab, avelumab) must be the most recent systemic anti-tumor treatment received in all patients, with documented progressive disease. Last administration of anti-PD-1 axis therapy must have been at least 3 weeks before the first dose of study drug.

a. Patients to be enrolled to the primary cohort (primary resistance) must have had progressive disease or stable disease less than 24 weeks as the best clinical response to anti-PD-1-axis monotherapy b. Patients to be enrolled to the exploratory cohort (acquired resistance) must have had stable disease for at least 24 weeks, partial response, or complete response as the best clinical response to anti-PD-1-axis monotherapy, with subsequent progression of disease J. At least one tumor amenable to incisional, excisional, core or forceps (transbronchial) biopsy. Patients must be willing to undergo tumor biopsies before starting trial therapy, and 9 to 10 weeks after initiation of therapy.

a. If the initial biopsy will be excisional, the excised tumor cannot be counted as a target lesion and there must be another lesion amenable to incisional, excisional, core or forceps biopsy. In this scenario, the second biopsy can only be excisional if the lesion to be excised is not a target lesion. b. Cytology tumor specimens (e.g. from fine-needle biopsies, or drainage of pleural/ pericardial or ascites fluid) are not acceptable. Biopsies of bone lesions that do not have a soft tissue component are also not acceptable (i.e. decalcified tumor samples are not acceptable).

K. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for 6 months after the last dose of trial therapy. Highly effective contraception is one with a failure rate of <0.1%. Birth control pills on their own do not achieve that rate.

1. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 72 hours of the start of study drug administration
2. Women who have recently given birth must no longer be breastfeeding

L. Adequate hematologic and end-organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment:

- Neutrophils ≥1500 cells/μL (without granulocyte colony-stimulating factor support within 2 weeks prior to Cycle 1, Day 1)

* Platelets ≥75,000/μL (transfusion to achieve this level is not permitted within 2 weeks of the first study drug administration)
* Hemoglobin ≥9.0 g/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x institutional upper limit of normal (ULN) with the following exceptions: Patients with documented liver metastases: AST and/or ALT≤5 x ULN
* Serum bilirubin ≤1.5 x ULN (Patients with known Gilbert disease who have serum bilirubin level ≤3 x ULN may be enrolled)
* Serum creatinine ≤1.5 x ULN or creatinine clearance ≥50 mL/min

Exclusion Criteria

A. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects who require intermittent use of inhaled steroids or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement, or psoriasis not requiring systemic therapy (within the past 3 years) will not be excluded from the study. B. Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity C. Subjects must not have a history of life-threatening toxicity related to prior anti-PD-1 axis therapy a. Subjects with history of anti-PD-1 axis therapy toxicities that are unlikely to recur with standard countermeasures (e.g., hormone replacement after adrenal crisis) are eligible.

D. Prior treatment with anti-CTLA-4 therapeutic antibodies

E. Symptomatic or untreated CNS metastases. Patients with a history of treated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

1. No evidence of interim progression between the completion of CNS-directed therapy and the start of trial therapy.
2. No ongoing requirement for dexamethasone as therapy for CNS disease; anticonvulsants at a stable dose are allowed.
3. Completed stereotactic radiosurgery at least 1 week prior to Cycle 1, Day 1 or wholebrain radiation at least 2 weeks prior to Cycle 1, Day 1 F. History of leptomeningeal carcinomatosis G. Prior palliative radiotherapy outside the CNS within 2 weeks of the first dose of study drug.

H. Treatment with systemic immunosuppressive medications (including but not limited to, dexamethasone at doses > 2 mg daily (or equivalent dose of other corticosteroids), cyclophosphamide, tacrolimus, sirolimus, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor [anti-TNF] agents) within 2 weeks prior to initiating trial therapy (Inhaled or topically applied steroids, and acute and chronic standard-dose NSAIDs are permitted. Replacement steroids are also permitted).

I. Subjects must not have received vaccines containing live virus for prevention of infectious diseases within 12 weeks prior to the first dose of study drug.

a. The use of inactivated seasonal influenza vaccines (eg, Fluzone®) will be permitted on study without restriction.

J. Any approved systemic anti-cancer therapy, within 3 weeks prior to initiation of study treatment; the following exception is allowed:

* TKIs approved for treatment of NSCLC discontinued > 7 days prior to Cycle 1, Day 1. The baseline scan must be obtained after discontinuation of prior TKIs.

K. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment; the following exceptions are allowed:

* Unapproved/experimental TKIs discontinued 14 days prior to Cycle 1, Day 1 L. Known infection with HIV, HBV or HCV. Patients with prior exposure to hepatitis, but no evidence of active or chronic infection, may be eligible.
* Subjects with positive hepatitis C antibody and negative quantitative hepatitis C by polymerase chain reaction are eligible.

M. Active systemic infection requiring systemic antibiotic treatment within 72 hours prior to first dose of study treatment N. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements O. Major surgery or traumatic injury within 4 weeks of starting study drug P. Women who are pregnant or lactating. Q. Any underlying medical condition that in the Principal Investigator's opinion will make the administration of study drug hazardous to the patient or would obscure the interpretation of adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Gettinger, M.D., Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Nivolumab and Ipilimumab - Primary | Combination Nivolumab and Ipilimumab - Acquired
Started | 10 | 10
Eligible for Biopsy | 7 | 7
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Nivolumab and Ipilimumab - Primary | Combination Nivolumab and Ipilimumab - Acquired | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 68.5 [54 to 76] | 64.5 [54 to 80] | 68.5 [54 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Using RECIST v1.1 to Nivolumab and Ipilimumab When Administered in Combination to Patients With Pre-treated Advanced NSCLC Who Have Experienced Primary Resistance to Anti-PD-1 Axis Therapy as Their Last Line of Systemic Therapy.
Description: Objective response is defined as a complete or partial response, as determined by investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 confirmed by repeat assessment ≥4 weeks after initial documentation. The categories are: complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD).
Time Frame: Tumor response assessment will occur every 9 weeks after initiating trial therapy for the first 24 weeks, and thereafter every 12 weeks until disease progression or up to 4 years.
Population: Patients that completed treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Nivolumab and Ipilimumab - Primary
Number analyzed (Participants) | 10
Participants
  complete response (CR) | 0
  partial response (PR) | 0
  stable disease (SD) | 2
  progressive disease (PD) | 8

2. Secondary Outcome: Objective Response Rate in in Advanced Non-small Cell Lung Cancer (NSCLC) With ACQUIRED Resistance to Anti-programmed Death (PD)-1 Axis Therapy as Their Last Line of Systemic Therapy.
Description: Objective response is defined as a complete or partial response, as determined by investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and confirmed by repeat assessment ≥4 weeks after initial documentation. The categories are: complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD). This outcome is only presented for those with advanced non-small cell lung cancer (NSCLC) with ACQUIRED resistance to anti-programmed death (PD)-1 axis therapy as their last line of systemic therapy.
Time Frame: Tumor response assessment will occur every 9 weeks after initiating trial therapy for the first 24 weeks, and thereafter every 12 weeks, up to four years.
Population: Patients with advanced non-small cell lung cancer (NSCLC) with ACQUIRED resistance to anti-programmed death (PD)-1 axis therapy as their last line of systemic therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Nivolumab and Ipilimumab - Acquired
Number analyzed (Participants) | 10
Participants
  complete response (CR) | 1
  partial response (PR) | 0
  stable disease (SD) | 8
  progressive disease (PD) | 1

3. Secondary Outcome: Progression-free Survival With Nivolumab and Ipilimumab When Administered in Combination to Patients With Pre- Treated Advanced NSCLC Who Have Experienced Primary Resistance to Anti-PD-1 Axis Therapy as Their Last Line of Systemic Therapy
Description: Progression free survival is defined as the time from the first day of nivolumab treatment until progression of disease using RECIST v1.1. This outcome is only presented for those pre-treated with advanced NSCLC who have experienced primary resistance to anti-PD-1 axis therapy as their last line of systemic therapy.
Time Frame: Until disease progression, unacceptable toxicity, or study termination, up to four years.
Population: Patients pre-treated with advanced NSCLC who have experienced primary resistance to anti-PD-1 axis therapy as their last line of systemic therapy.
Measure: Median (Full Range); unit: months
Arm/Group | Combination Nivolumab and Ipilimumab - Primary
Number analyzed (Participants) | 10
months | 1.8 [1.4 to 4.2]

4. Secondary Outcome: Progression Free Survival by RECIST v1.1 With Nivolumab and Ipilimumab in Patients With Pre-treated Advanced NSCLC Who Have Experienced Acquired Resistance to Anti-PD-1 Axis Therapy as Their Last Line of Systemic Therapy.
Description: Progression free survival is defined as the time from the first day of nivolumab treatment until progression of disease using RECIST v1.1 and immune related Response Criteria. This is in those that have experienced acquired resistance to anti-PD-1 axis therapy as their last line of systemic therapy.
Time Frame: Until disease progression, unacceptable toxicity, or study termination, up to four years from enrollment.
Population: Patients that completed treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Combination Nivolumab and Ipilimumab - Acquired
Number analyzed (Participants) | 10
months | 6.8 [1.8 to 28.7]

5. Secondary Outcome: Overall Survival (OS) With Nivolumab and Ipilimumab When Administered in Combination to Patients With Pre- Treated Advanced NSCLC Who Have Experienced PRIMARY Resistance to Anti-PD-1 Axis Therapy as Their Last Line of Systemic Therapy.
Description: Overall survival is defined as the time from the first day of treatment until death from any cause. If a patient has not experienced death, OS will be censored at the day of last follow-up. This is in patients that have experienced PRIMARY resistance to anti-PD-1 axis therapy as their last line of systemic therapy.
Time Frame: Until death or day of last follow-up, up to four years from enrollment.
Population: Patients that completed treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Combination Nivolumab and Ipilimumab - Primary
Number analyzed (Participants) | 10
months | 6.8 [1.7 to 17.8]

6. Secondary Outcome: Overall Survival With Nivolumab and Ipilimumab in Patients With Pre-treated Advanced NSCLC Who Have Experienced ACQUIRED Resistance to Anti-PD-1 Axis Therapy as Their Last Line of Systemic Therapy.
Description: Overall survival is defined as the time from the first day of treatment until death from any cause. If a patient has not experienced death, OS will be censored at the day of last follow-up.
Time Frame: Until death or day of last follow-up (up to four years from study enrollment).
Population: Patients that have completed treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Combination Nivolumab and Ipilimumab - Acquired
Number analyzed (Participants) | 10
months | 24.7 [7.5 to 48.5]

7. Secondary Outcome: Objective Response Rate Using irRC to Nivolumab and Ipilimumab When Administered in Combination to Patients With Pre-treated Advanced NSCLC Who Have Experienced PRIMARY or ACQUIRED Resistance to Anti-PD-1 Axis Therapy as Last Line of Systemic Therapy.
Description: Objective response is defined as a complete or partial response, as determined by investigator assessment using irRC and confirmed by repeat assessment ≥4 weeks after initial documentation.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Nivolumab and Ipilimumab - Primary | Combination Nivolumab and Ipilimumab - Acquired
Number analyzed (Participants) | 10 | 10
Participants | 0 | 1

8. Secondary Outcome: Safety of Nivolumab and Ipilimumab When Administered in Combination in Patients With Pre-treated Advanced NSCLC Who Have Experienced PRIMARY or ACQUIRED Resistance to Anti-PD-1 Axis Therapy as Their Last Line of Systemic Therapy.
Description: Determined based on adverse events which will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0. Presented are a count of those that experienced at least 1 Serious Adverse Event related to study drug.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Nivolumab and Ipilimumab - Primary | Combination Nivolumab and Ipilimumab - Acquired
Number analyzed (Participants) | 10 | 10
Participants | 2 | 2

9. Secondary Outcome: Feasibility of Sequential Biopsies in Patients With Pre-treated Advanced NSCLC Who Have Experienced PRIMARY or ACQUIRED Resistance to Anti-PD-1 Axis Therapy as Their Last Line of Systemic Therapy.
Description: Feasibility of sequential biopsies (performed or not performed) in patients with pre-treated advanced NSCLC who have experienced PRIMARY or ACQUIRED resistance to anti-PD-1 axis therapy as their last line of systemic therapy. Presented are a count of those that had biopsies performed or not performed.
Time Frame: Tumor biopsies performed at 9 to 10 weeks after receiving first dose of trial therapy.
Population: Only those that were eligible for biopsy at 9-10 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Nivolumab and Ipilimumab - Primary | Combination Nivolumab and Ipilimumab - Acquired
Number analyzed (Participants) | 7 | 7
Participants
  performed | 4 | 4
  not performed | 3 | 3

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Originally reported were deaths that occurred during treatment or within 30 days of treatment, the all cause mortality was updated to reflect a longer follow up time period.
Arm/Group | Combination Nivolumab and Ipilimumab - Primary | Combination Nivolumab and Ipilimumab - Acquired
All-Cause Mortality (participants affected / at risk) | 10/10 | 8/10
Serious Adverse Events (participants affected / at risk) | 3/10 | 2/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Nivolumab and Ipilimumab - Primary (N=10) | Combination Nivolumab and Ipilimumab - Acquired (N=10)
Autoimmune Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 1 (5)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 1 (1)
Parietal craniotomy (Surgical and medical procedures) | 0 (0) | 1 (2)
Radiation necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Nivolumab and Ipilimumab - Primary (N=10) | Combination Nivolumab and Ipilimumab - Acquired (N=10)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders -Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (8)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (4) | 4 (12)
General disorders - Other (General disorders) | 0 (0) | 2 (3)
Musculoskeletal and connective tissue disorders - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other (Eye disorders) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 1 (6)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 2 (3)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Hot Flashes (Vascular disorders) | 1 (1) | 0 (0)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 1 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03262779/Prot_SAP_000.pdf